CLINICAL TRIAL: NCT06571825
Title: Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation in Comparison to Consolidation Therapy Based Venetoclax for Elderly Patients With Acute Myeloid Leukemia After First CR
Brief Title: RIC Allo-HSCT vs. Venetoclax-Based Consolidation in Elderly AML Patients After First CR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Discipline Leader of Bone Marrow Transplant Center, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROPHY-AML03
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: elderly; AML; venetoclax; allo-HSCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Transplantation, Homologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAA group (Experimental)
  Interventions: Drug: Venetoclax
- HSCT group (Active Comparator)
  Interventions: Drug: Allogeneic transplant

INTERVENTIONS:
Drug: Venetoclax — The consolidation therapy involves a regimen of intermediate-dose cytarabine (Ara-C) combined with Ven, specifically Ara-C at 1.0 g/m²/day for 3 days (days 1-3) and Ven at 400 mg/day for 10 to 14 days (days 1-10 to 14), with each cycle lasting 4 to 6 weeks, for a total of 3 consolidation cycles. This is followed by maintenance therapy with azacitidine (AZA) at 50 mg/m²/day for 5 days (days 1-5), with each cycle lasting 4 weeks, for a total of 6 maintenance cycles.
  Arms: VAA group
Drug: Allogeneic transplant — The consolidation therapy involves allo-HSCT, with the choice of conditioning regimens typically using reduced-intensity conditioning such as the Fludarabine+Busulfan (FluBu) or Fludarabine+Melphalan (FluMel) regimens commonly used by centers, which can also include Ven.
  FluBu regimen: Flu 30 mg/m²/day from day -10 to day -5, Bu 3.2 mg/kg/day from day -6 to day -5 or day -7 to day -5, antithymocyte globulin (ATG) (e.g., rabbit ATG at a total dose of 6-7.5 mg/kg, administered from day -4 to day -1), and Ven from day -10 to day -4.
  FluMel regimen: Flu 30 mg/m²/day from day -10 to day -5, Mel 50-70 mg/m²/day from day -4 to day -3, ATG and Ven from day -10 to day -4.
  12 weeks (±4 weeks) post-HSCT maintenance begins with AZA at 32 mg/m²/day for 5 days (days 1-5), with each lasting 6 weeks, for a total of 6 cycles. Donor lymphocyte infusion is allowed in cases of minimal residual disease (MRD) positivity.
  Arms: HSCT group

SUMMARY:
Elderly patients with acute myeloid leukemia (AML) often face unfavorable prognostic factors such as multiple comorbidities, adverse cytogenetic profiles, and pre-existing hematological disorders. The long-term survival rate remains very low, with a 5-year survival rate of only 5% to 10%. The introduction of the BCL-2 inhibitor venetoclax (Ven) has improved the induction remission rates in elderly patients. However, the question of whether to use chemotherapy maintenance or proceed with allogeneic hematopoietic stem cell transplantation (allo-HSCT) for post-remission consolidation therapy remains unclear due to the lack of prospective controlled studies. Therefore, our center plans to conduct a prospective, open-label, two-arm, non-randomized, single-center study to further explore the optimal consolidation treatment strategy for elderly AML patients at intermediate and high risk following induction complete remission (CR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AML according to the 2022 WHO diagnostic criteria;
* Age 60-75 years;
* Intermediate to high-risk AML according to the ELN criteria, AML with myelodysplasia-related changes (AML-MRC) or therapy-related AML (t-AML), or core-binding factor AML (CBF-AML) with D816 KIT mutation; or newly diagnosed hypercellular leukemia (WBC ≥ 10×10^9/L);
* Achieved CR or CR with incomplete hematologic recovery (CRi) after one to two courses of induction chemotherapy;
* Have a matched related, haploidentical, or mismatched unrelated hematopoietic stem cell donor;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2; Creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula);
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3× the upper limit of normal (ULN), and total bilirubin ≤ 2× ULN;
* Echocardiography (ECHO) showing left ventricular ejection fraction (LVEF) ≥ 50%; Expected survival > 8 weeks;
* Voluntarily signed the informed consent form and can understand and comply with the study's requirements.

Exclusion Criteria:

* Currently has clinically active cardiovascular disease, such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, any class 3 or 4 heart disease according to the New York Heart Association (NYHA) functional classification, or a history of myocardial infarction within 3 months before screening;
* Other severe diseases that may limit the patient's participation in this trial (e.g., severe infection, renal failure);
* Known human immunodeficiency virus (HIV) infection or severe viral hepatitis not controlled by medication;
* Pregnant or breastfeeding women;
* Unable to understand, comply with the study protocol, or unable to sign the informed consent form.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | Up to 2 years
  Relapse-free survival (RFS) is measured from the date of achievement of first remission until the date of hematologic relapse or death from any cause.

SECONDARY OUTCOMES:
Non-Relapsed Mortality | Up to 2 years
  Non-relapsed mortality (NRM) is measured from the date of achievement of first remission until the date of death from any cause other than relapse.
Overall Survival | Up to 2 years
  OS is measured from the date of reaching CR1 to the date of death from any cause.
2-years Relapse Rate | Up to 2 years
  Relapse rate is defined as relapse probability at a given time point

OTHER OUTCOMES:
Minimal Residual Disease (MRD) Detected by Flow Cytometry | Up to 2 years
  Research on MRD involves using flow cytometry to detect residual cancer cells, with statistical methods including Kaplan-Meier survival analysis, Fine-Gray analysis and Cox regression modeling to evaluate disease remission and predict relapse risk.
Number of Participants With Treatment-Related Adverse Events (AEs) as Assessed by CTCAE v5.0 | Up to 2 years
  Research on AE uses descriptive statistics, Kaplan-Meier survival analysis, χ² or Fisher's exact tests to assess and compare AE incidence and survival outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Result] Kadia TM, Reville PK, Wang X, Rausch CR, Borthakur G, Pemmaraju N, Daver NG, DiNardo CD, Sasaki K, Issa GC, Ohanian M, Montalban-Bravo G, Short NJ, Jain N, Ferrajoli A, Bhalla KN, Jabbour E, Takahashi K, Malla R, Quagliato K, Kanagal-Shamanna R, Popat UR, Andreeff M, Garcia-Manero G, Konopleva MY, Ravandi F, Kantarjian HM. Phase II Study of Venetoclax Added to Cladribine Plus Low-Dose Cytarabine Alternating With 5-Azacitidine in Older Patients With Newly Diagnosed Acute Myeloid Leukemia. J Clin Oncol. 2022 Nov 20;40(33):3848-3857. doi: 10.1200/JCO.21.02823. Epub 2022 Jun 15. PMID 35704787
- [Result] Chua CC, Roberts AW, Reynolds J, Fong CY, Ting SB, Salmon JM, MacRaild S, Ivey A, Tiong IS, Fleming S, Brown FC, Loo S, Majewski IJ, Bohlander SK, Wei AH. Chemotherapy and Venetoclax in Elderly Acute Myeloid Leukemia Trial (CAVEAT): A Phase Ib Dose-Escalation Study of Venetoclax Combined With Modified Intensive Chemotherapy. J Clin Oncol. 2020 Oct 20;38(30):3506-3517. doi: 10.1200/JCO.20.00572. Epub 2020 Jul 20. PMID 32687450
- [Result] Wang H, Yao Y, Mao L, Lou Y, Ren Y, Ye X, Yang M, Ma L, Zhang Y, Zhou Y, Wu J, Huang X, Wang Y, Xu H, Tong H, Zhu HH, Jin J. Venetoclax plus '2 + 5' modified intensive chemotherapy with daunorubicin and cytarabine in fit elderly patients with untreated de novo acute myeloid leukaemia: a single-centre retrospective analysis. Br J Haematol. 2023 May;201(3):568-572. doi: 10.1111/bjh.18709. Epub 2023 Mar 2. No abstract available. PMID 36863709
- [Result] Garcia JS, Kim HT, Murdock HM, Cutler CS, Brock J, Gooptu M, Ho VT, Koreth J, Nikiforow S, Romee R, Shapiro R, Loschi F, Ryan J, Fell G, Karp HQ, Lucas F, Kim AS, Potter D, Mashaka T, Stone RM, DeAngelo DJ, Letai A, Lindsley RC, Soiffer RJ, Antin JH. Adding venetoclax to fludarabine/busulfan RIC transplant for high-risk MDS and AML is feasible, safe, and active. Blood Adv. 2021 Dec 28;5(24):5536-5545. doi: 10.1182/bloodadvances.2021005566. PMID 34614506